CLINICAL TRIAL: NCT04703530
Title: Effect of Hot Footbath on the Sleep Quality of Patients With Chronic Schizophrenia: A Randomized Controlled Trial
Brief Title: Effect of Hot Footbath on the Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Xuan-Yi Huang, RN, DNSc, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-108-05-176
Record Dates: First submitted 2020-09-25; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia
Keywords: Footbath; Quality of sleep; Chronic schizophrenia; Patient
MeSH Terms: conditions — Schizophrenia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The research was a randomized controlled trial. Participants were randomly allocated to the experimental group and the control group. The experimental group was given a hot footbath with a temperature of 41℃±1℃ for 20 minutes at about 1-2 hours before sleep, and this was repeated five times a week for four weeks; the control group was given routine care for four weeks. The CPSQI was used to collect the pre- and post-test data. Through this method, we explored whether the trial could effectively improve patients' sleep quality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot footbath effect on schizophrenia patient' sleep quality (Experimental): Participants were randomly allocated to the experimental group. The experimental group was given a hot footbath with a temperature of 41℃±1℃ for 20 minutes at about 1-2 hours before sleep, and this was repeated five times a week for four weeks. The CPSQI was used to collect the pre- and post-test data.
  Interventions: Other: hot footbath
- Routine care on schizophrenia patient' sleep quality (No Intervention): Participants were randomly allocated to the control group. They were given routine care for four weeks. The CPSQI was used to collect the pre- and post-test data.

INTERVENTIONS:
Other: hot footbath — The experimental group was given a hot footbath with a temperature of 41℃±1℃ for 20 minutes at about 1-2 hours before sleep
  Other Names: Experimental group
  Arms: Hot footbath effect on schizophrenia patient' sleep quality

SUMMARY:
The research title is the effect of hot footbath on the sleep quality of patients with chronic schizophrenia. The research was a randomized controlled trial. The setting was the chronic inpatient wards at a psychiatric teaching hospital in Northern Taiwan. A total of 63 participants, 30 in the hot footbath group and 33 in the control group, were completed the study from November 2019 to June 2020. Participants were randomly allocated to the experimental group and the control group. Through this method, we explored whether the trial could effectively improve patients' sleep quality.

DETAILED DESCRIPTION:
The research title is the effect of hot footbath on the sleep quality of patients with chronic schizophrenia. The research was a randomized controlled trial. The setting was the chronic inpatient wards at a psychiatric teaching hospital in Northern Taiwan. A total of 63 participants, 30 in the hot footbath group and 33 in the control group, were completed the study from November 2019 to June 2020. Participants were randomly allocated to the experimental group and the control group. The experimental group was given a hot footbath with a temperature of 41℃±1℃ for 20 minutes at about 1-2 hours before sleep, and this was repeated five times a week for four weeks; the control group was given routine care for four weeks. The CPSQI was used to collect the pre- and post-test data. Through this method, we explored whether the trial could effectively improve patients' sleep quality.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Schizophrenia Disease.
2. Having Schizophrenia at least two years.
3. Must have above 5 scores in the Pittsburgh Sleep Quality Index (CPSQI).

Exclusion Criteria:

1. Having the foot problems, including allergy, wound, swelling, pain, peripheral circulation, and any skeletal, muscular, or nervous lesions in the foot.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | pretest
  index scoring from 0 to 3 points, and total 21 points. A total score of all seven indexes > 5 suggests poor sleep quality
Pittsburgh Sleep Quality Index | up to 4 weeks
  index scoring from 0 to 3 points, and total 21 points. A total score of all seven indexes > 5 suggests poor sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Xuan-Yi Huang, DNSc, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- Tri-Service General Hospital Beitou Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan MS, Chung KF, Yung KP, Yeung WF. Sleep in schizophrenia: A systematic review and meta-analysis of polysomnographic findings in case-control studies. Sleep Med Rev. 2017 Apr;32:69-84. doi: 10.1016/j.smrv.2016.03.001. Epub 2016 Mar 10. PMID 27061476
- [Result] Seyyedrasooli A, Valizadeh L, Zamanzadeh V, Nasiri K, Kalantri H. The effect of footbath on sleep quality of the elderly: a blinded randomized clinical trial. J Caring Sci. 2013 Nov 30;2(4):305-11. doi: 10.5681/jcs.2013.036. eCollection 2013 Dec. PMID 25276739
- [Result] Sung EJ, Tochihara Y. Effects of bathing and hot footbath on sleep in winter. J Physiol Anthropol Appl Human Sci. 2000 Jan;19(1):21-7. doi: 10.2114/jpa.19.21. PMID 10979246
- [Result] Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res. 2005 Oct;14(8):1943-52. doi: 10.1007/s11136-005-4346-x. PMID 16155782
- [Result] Valizadeh L, Seyyedrasooli A, Zamanazadeh V, Nasiri K. Comparing the Effects of Reflexology and Footbath on Sleep Quality in the Elderly: A Controlled Clinical Trial. Iran Red Crescent Med J. 2015 Nov 1;17(11):e20111. doi: 10.5812/ircmj.20111. eCollection 2015 Nov. PMID 26734475
- [Result] Yang HL, Chen XP, Lee KC, Fang FF, Chao YF. The effects of warm-water footbath on relieving fatigue and insomnia of the gynecologic cancer patients on chemotherapy. Cancer Nurs. 2010 Nov-Dec;33(6):454-60. doi: 10.1097/NCC.0b013e3181d761c1. PMID 20562619
- See also: Sleep in schizophrenia: A systematic review and meta-analysis of polysomnographic findings in case-control studies. Sleep Medicine Reviews, 32, 69-84. — https://pubmed.ncbi.nlm.nih.gov/27061476/
- See also: Effects of bathing and hot footbath on sleep in winter — https://doi.org/10.2114/jpa.19.21
- See also: Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control Subjects — https://doi.org/10.1007/s11136-005-4346-x
- See also: Comparing the effects of reflexology and footbath on sleep quality in the elderly: A controlled clinical trial — https://doi.org/10.5812/ircmj
- See also: The Effects of Warm-Water Footbath on Relieving Fatigue and Insomnia of the Gynecologic Cancer Patients on Chemotherapy — https://doi.org/10.1097/ncc.0b013e3181d761c1